CLINICAL TRIAL: NCT06143813
Title: Precision Treatment of Lumbar Spine Surgery Through Advanced Nerve Root Blockade
Acronym: PLAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Private Hospital Moelholm (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PLAN
Record Dates: First submitted 2023-11-09; First posted 2023-11-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2023-11

CONDITIONS: Radiculopathy Lumbar; Radiculopathy Sacral; Herniated Disc; Foraminal Stenosis; Stenosis, Spinal
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Block (Active Comparator): This group will receive standard of care + a selective nerve root block as part of the diagnostic work up.
  Interventions: Diagnostic Test: Selective nerve root block (SNRB)
- No-block (No Intervention): This group will receive standard of care.

INTERVENTIONS:
Diagnostic Test: Selective nerve root block (SNRB) — CT/Fluoroscopy guided nerve root block
  Other Names: Transforaminal nerve root block
  Arms: Block

SUMMARY:
The overall purpose of the study is to investigate whether selective spinal nerve root blocks can improve diagnostics of radiculopathy due to lumbar disc herniation (LDH), foraminal stenosis (FS), and recess stenosis (RS), and hence identify the patients that will benefit from surgical intervention.

DETAILED DESCRIPTION:
The study is designed as a prospective randomized controlled trial, using a two-group stratified block-randomization, evaluating the effect of adding the outcome of a diagnostic SNRB to surgical decision-making. Stratification will be based on the study site. Block size will be 4, 6, or 8 and in random order.

All patients referred to our departments with suspected radiculopathy and radiological evidence of root compression are eligible for inclusion. Patients will be randomized to either standard care or SNRB after the consultation. Results of the SNRB will be available to the surgeon before deciding finally whether to operate or not. Hence, the intervention adds the outcome of the diagnostic SNRB to the shared surgical decision-making.

Study outline:

Baseline:

Demographics, Oswestry Disability Index, Eq5D, SF-36, NRS-LP, and NRS-BP will be recorded

1-month follow-up after surgery: Oswestry Disability Index, Eq5D, SF-36, NRS-LP, and NRS-BP will be recorded

3-months follow-up after surgery: Oswestry Disability Index, Eq5D, SF-36, NRS-LP, and NRS-BP will be recorded

12-months follow-up after surgery: Oswestry Disability Index, Eq5D, SF-36, NRS-LP, and NRS-BP will be recorded

Randomization:

Using RedCap patients will be randomized to receive a SNRB as part of the pre-operative workup or to direct operation.

SNRB-procedure:

At Aarhus University, the SNRB will be performed using CT-guidance; at Private Hospital Moelholm, the SNRB procedure will be guided by fluoroscopy. Drugs used are omnipaque (0,2 ml), betamethasone (0,5 ml) and bupivacain (0,5 ml)

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Suspected lumbar radiculopathy persistent ≥ 8 weeks
* Radiological evidence of lumbar nerve root compression (herniated disc, recess stenosis, foraminal stenosis)

Exclusion Criteria:

* Prior lumbar spine surgery
* Mental illness
* Language barrier in Danish
* Severe physical co-morbidity
* Known allergies to medicine used in the study
* Pregnant
* Plans to move abroad during the next 12-months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Minimum clinically important difference (MCID) | 3 months after surgery/decision not to operate
  Difference in mean change on numerical rating scale for leg pain (NRS-LP) 3 months after surgery. The margin of non-inferiority will be set to = 1.6 points. Comparison will be made between patients in the SNRB group and patients in the control group surgery.

SECONDARY OUTCOMES:
Leg pain | 3 months after surgery/decision not to operate
  Difference in proportions reaching 1.6 points on NRS-LP 3 months after surgery/decision to not to operate. Comparison will be made between the SNRB group and the standard of care group.
Back pain | 3 months after surgery/decision not to operate
  Mean change in numerical rating scale for back pain (NRS-BP) 3 months after surgery/decision to not to operate. Comparison will be made between the SNRB group and the standard of care group.
SF-36 (Short form 36) | 3 months after surgery/decision not to operate
  SF-36 3 months after surgery/decision to not to operate. Comparison will be made between the SNRB group and the standard of care group.
EQ5D (EuroQol 5D) | 3 months after surgery/decision not to operate
  EQ5D 3 months after surgery/decision to not to operate. Comparison will be made between the SNRB group and the standard of care group.
ODI | 3 months after surgery/decision not to operate
  Oswestry Disability Index (ODI) 3 months after surgery/decision to not to operate. Comparison will be made between the SNRB group and the standard of care group.
Subanalysis | 3 months after surgery
  Fraction of patients not reaching minimum clinically important difference (MCID) on the numerical rating scale for leg pain (NRS-LP) 3 months after surgery (MCID NRS-LP = 1.6 points). Comparison will be made between patients in the SNRB group who underwent surgery and patients in the control group that underwent surgery.

CONTACTS AND LOCATIONS:
Overall Officials: David Kocemba, MD, Principal Investigator — University of Aarhus; Mikkel Rasmussen, MD, Study Director — University of Aarhus; Bent Uhrbrand, MD, Study Chair — Private Hospital Moelholm
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kocemba D, Andersen PA, Carlsen JG, Schulz MK, Uhrbrand B, Dinesen H, Mikkelsen R, Thygesen M, Rasmussen MM. The PLAN trial: precision treatment of lumbar spine surgery with advanced nerve root blockade - protocol for a prospective, investigator-initiated, randomized non-inferiority trial. BMC Musculoskelet Disord. 2025 Dec 12. doi: 10.1186/s12891-025-09395-0. Online ahead of print. PMID 41388268